CLINICAL TRIAL: NCT00213629
Title: Transcriptome Analysis Through a Dedicated Macro-array and TcLandscape Repertoire Analysis for Diagnosis of Myositis.
Brief Title: myoARRAY and TcLandscape Analysis for the Diagnosis of Inflammatory Myopathies
Acronym: MYOARRAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2003/094/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Polymyositis; Dermatomyositis
Keywords: myositis; cDNA arrays; Genes, T-Cell Receptor beta
MeSH Terms: conditions — Polymyositis; Dermatomyositis; Myositis | interventions — Gene Expression Profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- no arm (Other): no arm
  Interventions: Other: transcriptome analysis; Other: T cell repertoire analysis

INTERVENTIONS:
Other: transcriptome analysis — transcriptome analysis from muscle biopsy
Other: T cell repertoire analysis — blood T cell repertoire analysis

SUMMARY:
The diagnosis of the different forms of inflammatory myopathies (polymyositis, dermatomyositis, inclusion-body myositis...) remains difficult which may lead to unappropriate patient care.

Objective 1 : to develop and evaluate the diagnostic value of a dedicated DNA-array (myoARRAY) for adult-onset muscular diseases with focus on inflammatory myopathies.

Objective 2 : to evaluate the diagnostic value of T cell repertoire (TcLand) analysis to distinguish different forms of inflammatory myopathies.

ELIGIBILITY:
Inclusion Criteria:

* indication of muscle biopsy for diagnostic purpose
* written informed consent

Exclusion Criteria:

* vasculitis
* coagulation disorder, impossibility to perform muscle biopsy

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
transcriptome | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Boyer, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- University Hospital of Rouen, Rouen, Seine Maritime, France